CLINICAL TRIAL: NCT02977702
Title: Sarcopenia is an Independent Prognostic Factor for Overall Survival in Patients With Pancreatic Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Other Study IDs: ICL_2015_0003
Record Dates: First submitted 2016-11-28; First posted 2016-11-30 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
The primary objective of this study was to validate Total Psoas Area (TPA) measurement as an independent prognostic factor of overall survival in patients with pancreatic adenocarcinoma. Secondary objective was to describe the evolution of the TPA during the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* All patients consecutive enrolled from January 2009 to December 2015 who underwent at least one chemotherapy for pancreatic adenocarcinoma, whatever the stage

Exclusion Criteria:

* A patient record captured outside the time frame from January 2009 to December 2015

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients records would be extracted from the electronic health record system of Institut de Cancérologie de Lorraine
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2015-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
overall survival | 24 months